CLINICAL TRIAL: NCT05236387
Title: A Single-Center, Open-Label Study Evaluating the Ability of 99mTc-Tilmanocept to Identify Clipped Nodes in Breast Cancer Patients Undergoing Neoadjuvant Chemotherapy and Sentinel Lymph Node Dissection
Brief Title: Evaluating the Ability of 99mTc-Tilmanocept to Identify Clipped Nodes in Breast Cancer Patients Undergoing Neoadjuvant Chemotherapy and Sentinel Lymph Node Dissection
Status: Terminated | Type: Observational
Why Stopped: PI left institution
Sponsor: Johns Hopkins University (Other)
Collaborators: Cardinal Health (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB00154162
Record Dates: First submitted 2022-01-18; First posted 2022-02-11 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
Keywords: Lymphoseek; Sentinel Lymph Nodes; Neo Adjuvant Chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — technetium Tc 99m tetramethyl-propyleneamine oxime; technetium-diethylenetriaminepentaacetic acid-mannosyl-dextran

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intent to Treat group: All patients meeting entrance criteria, injected with 99m Tc-TM, and having one or more lymph nodes removed for which the pathologist confirms the type (lymph node versus non-lymph node) and contents (e.g., tumor cells) of the excised tissues will comprise the intent-to-treat population (ITT). This definition also carries over to the lymph nodes; i.e., nodes used for the ITT analysis must come from patients included in the ITT population. The ITT population will serve as the analysis population for all efficacy endpoints, unless indicated otherwise in the description of analyses.
  Interventions: Drug: 99m Tc-TM

INTERVENTIONS:
Drug: 99m Tc-TM — Each patient will receive a single injection (0.1 ml) of 99mTc-TM (50 mcg) at the upper outer skin of the breast using an intradermal technique confirmed by the presence of a skin wheal.
  Other Names: Lymphoseek

SUMMARY:
The purpose of the present study is to evaluate the ability of 99mTc-TM to identify the clipped node after neoadjuvant chemotherapy (NAC) and to compare this percentage with historical national data. This study will also evaluate pain and discomfort after injection and pathological features of clipped nodes and any additional nodes removed.

DETAILED DESCRIPTION:
This is a phase 4 single-center, open-label, single-arm study evaluating the ability of 99mTc-TM to identify clipped nodes in primary breast cancer patients receiving NAC and subsequent Sentinel Lymph Node Biopsy (SLNB) as practice compared to published historical data . Sixty-four (64) patients (≥18 years) diagnosed with breast cancer and who are evaluated as having a favorable response (i.e., at least partial clinical response in the breast) to chemotherapy during the mid-treatment evaluation will be evaluated in this study. Patients will have suspicious lymph nodes assessed and one biopsied for pathological evaluation and clipped during the course of the patients' medical work-up. Patients will undergo NAC treatment and have a mid-treatment evaluation to assess response to the chemotherapy. Patients with a favorable response will complete NAC followed by identification of the clipped node and sentinel lymph nodes and standard lymph node assessment. Patients with an unfavorable response (i.e., no response to the NAC) will continue NAC but will not continue to participate in the study. All study patients undergoing SLNB will receive a single injection (0.1 ml) of 99mTc-TM (50 mcg) preoperatively. If no signal is detected within 30-60 minutes, patients may also be injected with BD (up to 10 cc), intraoperatively. Pain at injection site will be assessed pre-injection and at 1 minute after the 99mTc-TM injection.

It is anticipated that the majority of patients enrolled will receive NAC treatment. Although chemotherapy will be the primary neoadjuvant treatment used in this study, if the investigator feels the patient will benefit more from hormonal therapy, a hormonal treatment will be administered.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has provided written informed consent with HIPAA authorization.
2. The patient is female or male and ≥18 years of age at the time of consent.
3. The patient has been diagnosed with invasive Stage 2-3 breast cancer (T1-3; N1-2).
4. The patient has no history of inflammatory breast cancer.
5. The patient has no matted node on examination (N3).
6. The patient is eligible for neoadjuvant chemotherapy (NAC).
7. The patient is a candidate for surgical intervention, with sentinel lymph node assessment being a part of the surgical plan.
8. If of childbearing potential, the patient has a negative pregnancy test within 48 hours before administration of Lymphoseek, has been surgically sterilized, or has been postmenopausal for at least 1 year.
9. The patient has no known allergies or hypersensitivity to 99mTc-TM, BD, or India ink.

Exclusion Criteria:

1. The patient is pregnant or lactating.
2. The patient has clinical and/or radiological evidence of metastatic or systemic disease. Oligo metastatic disease is acceptable (one organ and controlled).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intent-to-treat population All patients meeting entrance criteria, injected with 99mTc-TM, and having one or more lymph nodes removed for which the pathologist confirms the type (lymph node versus non-lymph node) and contents (e.g., tumor cells) of the excised tissues will comprise the intent-to-treat population (ITT). This definition also carries over to the lymph nodes; i.e., nodes used for the ITT analysis must come from patients included in the ITT population. The ITT population will serve as the analysis population for all efficacy endpoints, unless indicated otherwise in the description of analyses.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Percentage of clipped nodes detected with 99m Tc-Tm intraoperatively as determined with a hand held gamma detection device | 1 month after the surgery
  The percentage of clipped nodes identified using 99mTc-TM will be calculated, along with an exact binomial 95% confidence interval.

SECONDARY OUTCOMES:
Change in Pain at injection site as assessed by a visual analog scale | Immediately before injection and at 1 minute after injection
  Pain Assessment will be performed before injecting 99m Tc-TM and approximately 1 minute after the injection. Injection site pain will be assessed using a standardized visual analog scale (VAS). The VAS is a horizontal line measuring 0-100 mm in length, anchored by word descriptors at each end. The left end (0 mm) is labeled "no pain" and the right end (100 mm) is labeled "worst pain imaginable". The patient will be instructed to make a vertical mark on the horizontal line that they feel represents their pain intensity. The VAS is scored manually by measurement in millimeters from the left side of the line (0 mm) to the point where the patient marks on the horizontal line.
Number of clipped nodes that were SLNs | 1 month after the surgery
  Number of clipped nodes that were Sentinel Lymph Nodes (SLNs).
Concordance of blue/hot nodes for clipped and SLNs as assessed by Lymphoseek with the highest counts on the Gamma counter | 1 month after the surgery
  To study the pathological features of the clipped node and any additional nodes (attempt for 2-3 total sentinel lymph node assessment, as standard practice) identified by Lymphoseek with the highest counts on the Gamma counter (10% rule).

CONTACTS AND LOCATIONS:
Overall Officials: Mehran Habibi, MD, Principal Investigator — Johns Hopkins Bayview
Locations (1):
- Johns Hopkins Bayview Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No